CLINICAL TRIAL: NCT01392287
Title: Treatment Resistant Geriatric Depression in Primary Care: Is NAAG (N-Acetylaspartylglutamate), Measured by Proton Magnetic Resonance Spectroscopy (1H-MRS) at 3 Tesla, a Predictor of Treatment Response?
Brief Title: Treatment Resistant Geriatric Depression in Primary Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Cambridge Health Alliance (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Brent Forester, Geriatric Psychiatrist / Principal Investigator, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-P-001094
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Major Depressive Disorder
Keywords: Geriatric; Older adults; Major Depressive Disorder; Magnetic Resonance Spectroscopy; memantine hydrochloride; N-Acetylaspartylglutamate; NAAG; Cognitive impairment
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine hydrochloride (Experimental): Older individuals with DSM IV TR Major Depression, with persistent symptoms of depression despite at least 8 weeks of treatment with standard pharmacotherapy, will be referred for a study of memantine hydrochloride augmentation. Healthy control subjects follow similar study schedule for baseline and endpoint but do not receive memantine hydrochloride.
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Dosing Form: Tablet
  Dosage: 5mg, 10 mg
  Description:
  Memantine hydrochloride (Namenda®), a low to moderate affinity uncompetitive (open-channel) NMDA antagonist, is manufactured and supplied by Forest Laboratories, Incorporated. Only the subjects in the depression group will receive the study drug memantine HCl. Per psychiatrist's instructions, subjects may remain on the maximum dosage of memantine HCl allowed by the study protocol for a given week, or reduce the dosage if concerns regarding tolerability arise. The dosage of memantine HCl cannot be increased more rapidly than the dosing schedule listed below.
  Memantine HCl Dosing Schedule:
  5 mg qAM week 1 5 mg qAM and 5 mg qHS for week 2 10 mg qAM and 5 mg qHS for week 3 10 mg BID for week 4, 5, 6, 7, and 8
  Other Names: Namenda (NDA # 021487)

SUMMARY:
This study involves collaboration between McLean Hospital, Geriatric Medicine at the Cambridge Health Alliance (CHA) and other sites within the Partners and Harvard Medical School network. The investigators plan to recruit individuals 55 to 89 years old with treatment resistant depression. Someone with "treatment resistant" depression for this study may be someone who still has sad or low feelings and thoughts even though he/she is taking an antidepressant medication for at least 8 weeks to help relieve his/her depression. During the study, subjects will gradually add memantine hydrochloride in dosages up to 20 mg/day for 8 weeks to their standard antidepressant treatment.

The investigators are doing this research study to help answer 3 questions:

1. Do older adults with treatment resistant Major Depression have lower levels of a chemical in the brain called NAAG than older adults without Major Depression?
2. Do older adults with naturally low NAAG levels do better on memantine hydrochloride treatment than older adults with higher amounts of this chemical on memantine hydrochloride treatment?
3. Do older adults with treatment resistant depression have more problems with memory and concentration than older adults without depression?

The investigators are also interested in looking at electrical and neuronal activity of the brain, spiritual beliefs, and fatigue in relationship to depression.

The investigators hypothesize that:

1. Older individuals with treatment resistant Major Depression will have lower levels of NAAG compared with age-matched older control subjects.
2. Older adults with treatment resistant depression and low NAAG levels will do better on treatment with memantine hydrochloride than older adults on memantine with higher NAAG levels.
3. Older adults with depression will do better on tests of attention and executive functioning after treatment with memantine hydrochloride.
4. Healthy controls will do better on tests of attention and executive functioning than older adults with depression.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS

We will enroll up to 20 subjects with major depression, ages 55-89, and up to 20 healthy control subjects, ages 55-89 matched with depression group for age, sex, and ethnicity. We require 10 subjects in each group to have completed the study protocol with clinical and MRI scan data suitable for analysis.

Subjects in both groups will be recruited from:

* Cambridge Health Alliance (CHA) geriatric medicine group practice.
* Mount Auburn Outpatient programs and affiliates
* Beth Israel Deaconess Medical Center Outpatient programs and affiliates
* McLean Hospital Geriatric Psychiatry Outpatient, Inpatient, and Partial (SAGE - Seniors Aging Gracefully Everyday) programs
* Other inpatient, partial, and outpatient psychiatry programs at McLean Hospital
* Outpatient programs affiliated with Partners Healthcare and/or Harvard Medical School, such as:
* Partners Community Health Care primary care physicians (PCPs),
* Massachusetts General Hospital and Brigham and Women's PCP network
* Local geriatricians and community psychiatrists
* General public and community (through IRB-approved local advertisements), such as:
* Public areas (gyms, super markets, etc)
* Retirement communities
* The Harvard Division on Aging
* Newspaper
* Radio
* Internet
* McLean Hospital Geriatric Psychiatry Research Program's research studies, including:
* Subjects who have completed participation in treatment or non-treatment studies
* Subjects who are actively participating in non-treatment research studies

One site (McLean Hospital) is engaged in this protocol. CHA and other sites only refer subjects to McLean and do not consent subjects or complete any study protocol procedures. Subjects must meet all selection criteria in order to participate in the study protocol.

All subjects will complete a brief pre-screening interview over the phone or in person in order to assess their preliminary eligibility for study inclusion.

Screening Period:

After signing consent, all study subjects will follow the same screening period (with the exceptions for control subjects mentioned below). Screening procedures include a clinical diagnostic interview, medical monitoring, physical exam, collecting information regarding prior and concomitant medication and adverse events, blood draw, vital signs, height, and weight, demographic and clinical history information, as well as assessments of daily functioning, mood, anxiety, and cognition.

Visit 2 / Baseline (Week 0):

Depression subjects will return to the office after the completion of screening procedures (within 14 days of signing consent) to complete baseline procedures which include assessments of daily functioning, fatigue, mood, anxiety, medical monitoring, psychiatric interview, concomitant medications, adverse events, vitals, 3T scan, EEG with resting state and Flanker Task procedures (prior to receiving study medication), spirituality questionnaire, and urine pregnancy test (if applicable). Neuropsychological tests will also be completed at this visit.

No changes in psychotropic drugs will be allowed for depression subjects during this the screening period before study drug is administered. The subjects with depression will be administered (before leaving the office) memantine HCl 5 mg tablets. All depression subjects will start at a dose of 5 mg once per day in the morning.

Visit 3 (Week 1) and Visit 4 (Week 2):

Following the completion of Visit 2, the subject will return to the office for 2 visits in 2 consecutive weeks. A psychiatric interview, review concomitant medications and AEs (if any), mood and anxiety scales, monitoring of medication tolerability and compliance, vital sign collection will be completed at these visits. Study medication will be dispensed and depression subjects will be instructed according to the dosing schedule.

Visit 5 (Week 4) and 6 (Week 6):

After completing Visit 4, subjects will return to the office 2 weeks later for Visit 5 (Week 4) and then 2 weeks after that for Visit 6 (Week 6). The same visit procedures will be completed at these visits as Visits 3 and 4, except the subject will not meet with the study psychiatrist at Visit 6 (Week 6). Subjects may complete Visit 6 in person or over the phone.

Visit 7 (Week 8) Final Study Visit:

After completing 8 weeks on study medication, the subject will return to the office for the final study visit. This visit will complete the same procedures as Visits 3 through 6 with the addition of another 3T scan (with a negative urine pregnancy test, if applicable), EEG (with resting state and Flanker Task) and neuropsychological tests. Participants will also repeat spirituality and fatigue questionnaires with assistance from study staff.

Subjects will be asked to return all study medication for the final visit. At this time subjects will have the option of staying on the medication or tapering off study medication and being referred to the McLean Hospital Geriatric Outpatient Clinic for follow up or to an appropriate physician of their choice. We will share information regarding study participation and results with the subjects' primary care physician and/or other entities only if the subject has completed an "Authorization for Release of Medical Records" form. If the subjects chose to discontinue treatment with memantine HCl, the psychiatrist (BPF) will instruct subjects how to safely taper off study medication.

Control Subject Visits:

Following screening, control subjects will return to the office for 3 visits. Unlike the depression group, the control group will NOT receive the study drug memantine HCl. Control subjects are not scheduled to meet with the study psychiatrist at the Baseline Week 0 and Week 8 visits and complete blood draw and one of the neuropsychological tests during participation. Other than the exceptions previously mentioned, control subjects will follow the same protocol as the depression subjects for the screening period, Baseline (Week 0), and Week 8 Visit. Study staff will monitor adverse events (if any occur), use of concomitant medication (if any), and subject safety throughout study participation. Vital signs will also be collected at every visit. Mood measures, spirituality and fatigue questionnaires, and neuropsychological tests identical to those administered to the depression group will be completed during the Week 8 final visit. Controls will also complete the same 3T MRI scanning protocol as depression subjects. Controls also have the opportunity to participate in EEG acquisition at baseline and study endpoint.

Follow-up:

We plan to contact enrolled subjects after the last subject completes the study per protocol and the data has been analyzed. This follow-up correspondence will consist of at least 3 attempts to contact subjects' by phone and 1 certified letter sharing our research findings with subjects.

ELIGIBILITY:
Inclusion Criteria for Depression Subjects:

* Ability to provide informed consent
* Age 55 to 89, inclusive
* DSM-IV Diagnosis of Major Depressive Disorder
* MADRS score of >16 at screening and baseline*
* Must speak, read, and write in English
* On standard antidepressant medication for at least 8 weeks prior to beginning memantine hydrochloride treatment

Exclusion Criteria for Depression Subjects:

* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder
* History or current diagnosis of the following psychiatric illnesses: any organic mental disorder (including dementia), schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specified, bipolar disorder, patients with substance dependence disorders, including alcohol, active within the last 12 months
* History of drug hypersensitivity or intolerance to memantine hydrochloride
* Use of the following class of medications: barbiturates.**
* Inability to complete the screening procedures
* Contraindications to magnetic resonance imagining (MRI), including any of the exclusion criteria mentioned in the MRI risks section of this protocol
* MRI abnormality that compromises integrity of imaging data (eg. intracranial lesions, hydrocephalus)
* Non-English speaking participants

Notes for Study Criteria (Depressed Subjects):

*Depressed subjects that score below a 16 on the MADRS at baseline may be reevaluated within two weeks. After reevaluation, study staff will exclude subjects that continue to score below a 16 on the MADRS. All subjects who score 16 or above at reevaluation may be included in the study at that point, provided they still meet study criteria.

**Benzodiazepines and non-benzodiazepine sedative hypnotics (such as zolpidem/Ambien), may be used by depressed subjects throughout the study as long as they are not taken within 12 hours of any MRI scan.

Inclusion Criteria for Control Subjects:

* Ability to provide informed consent
* Age 55 to 89, inclusive
* MADRS score <4
* Must speak, read, and write in English
* Must match with a depression subject previously enrolled on age (+/- 5 years) and sex

Exclusion Criteria for Control Subjects:

* Any evidence of current or past psychiatric disorders
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder
* History or current diagnosis of the following psychiatric illnesses: any organic mental disorder (including dementia), major depressive disorder, depression NOS, dysthymia, bipolar disorder( type I or II), schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specified, bipolar major depressive disorder, patients with substance dependence disorders, including alcohol.
* Use of any class of psychotropic medication.
* Inability to complete the screening visit
* MRI abnormality that compromises integrity of imaging data
* Contraindications to magnetic resonance imagining (MRI), including any of the exclusion criteria mentioned in the MRI risks section of this protocol
* Non-English speaking participants

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mean Differences in NAAG Levels between Subject Groups at Baseline and Week 8 | Baseline / Study Entry
  Are NAAG levels are lower in older adults with treatment resistant depression compared with healthy age-matched controls?

SECONDARY OUTCOMES:
Relationship of NAAG Levels and MADRS Scores between Subject Groups at Baseline and Week 8 | 8-week trial
  Do subjects with low NAAG levels within the treatment resistant depression group prior to memantine hydrochloride augmentation respond better to treatment with memantine hydrochloride?
Cognitive Impairment between Subject Groups at Baseline and Week 8 | 8-week trial
  Do older adults with Major Depression have evidence of cognitive impairment (in particular in the realm of executive functioning and attention) compared with older healthy controls from baseline to study endpoint?

CONTACTS AND LOCATIONS:
Overall Officials: Brent P Forester, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Harvard Catalyst Website — http://catalyst.harvard.edu/